CLINICAL TRIAL: NCT01095783
Title: Treatment of Low Back Pain in Patients With End-stage Renal Disease on Hemodialysis
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: My main collaborator got sick and cannot continue the project. The study ended.
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Ricardo de Castro Cintra Sesso, Associate Professor, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CEP 0087/09; cep 0087/09 (Other: Federal University of São Paulo)
Record Dates: First submitted 2010-03-29; First posted 2010-03-30 (Estimated); Last update posted 2015-08-11 (Estimated); Status verified 2015-08

CONDITIONS: Chronic Low Back Pain
Keywords: low back pain; physiotherapy; hemodialysis; end-stage renal disease
MeSH Terms: conditions — Low Back Pain; Kidney Failure, Chronic

ARMS (2):
- Physiotherapeutic intervention (Experimental)
  Interventions: Procedure: physiotherapeutic intervention
- control (Other): The control group receive transcutaneous electrical nerve stimulation (TENS) for 20 min at 50-100 Hz frequencies for the same time frame (Anesth Analg 2004;98:1552-6)
  Interventions: Procedure: control

INTERVENTIONS:
Procedure: physiotherapeutic intervention — Twenty repetitive exercises (30 seconds per exercise) consisting of: flexion in standing, extension in standing, flexion in lying, and extension in lying position applied three times a week for eight weeks
  Arms: Physiotherapeutic intervention
Procedure: control — The control group receive transcutaneous electrical nerve stimulation (TENS) for 20 min at 50-100 Hz frequencies for the same time frame (Anesth Analg 2004;98:1552-6)
  Arms: control

SUMMARY:
The purpose of this study is to determine whether a physiotherapeutic intervention is effective in the treatment of low back pain in hemodialysis patients

DETAILED DESCRIPTION:
Low back pain is a significant morbidity in chronic hemodialysis patients affecting about 1/3 of them. Among the physiotherapeutic interventions, the McKenzie Method (Spine 1983;8:141-4), has shown to be an effective approach to manage patients with low back pain. More specifically, it consists on standardized repetitive flexion and extension exercises of the lumbar spine. Thus far, there has been no randomized intervention testing the effectiveness of physiotherapeutic interventions in chronic renal failure patients on hemodialysis. In this study we selected four of their main proposed exercises (flexion in standing, extension in standing, flexion in lying, and extension in lying position) to apply three times a week for eight weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic low back pain
* Chronic renal failure
* Hemodialysis therapy for more than 3 months

Exclusion Criteria:

* Fractures of the spine
* Psychiatric diseases
* Alcohol of other drugs use
* Planned living donor transplantation
* Clinically unstable patients
* Chronic neurologic diseases

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-03; Primary Completion 2013-09 (Estimated); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
Improvement in functional status of the lumbar spine as measured by the Roland Morris Disability questionnaire, consisting of 24 items wich are reported by the patient. Additionally, the lumbar pain will be assessed by a visual analogue scale. | eight weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Federal University of São Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Cristofolini T, Draibe S, Sesso R. Evaluation of factors associated with chronic low back pain in hemodialysis patients. Nephron Clin Pract. 2008;108(4):c249-55. doi: 10.1159/000124328. Epub 2008 Apr 9. PMID 18401192